CLINICAL TRIAL: NCT03618615
Title: Anatomical Study of the Arteries of the Skin on Amputation Legs
Acronym: APIA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02936-47
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Arteritic Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial patient coming to CHRU Nancy, in the Vascular and Endoluminal Surgery Department, to undergo leg amputation.
  Usually, after the amputation of the leg in the operating theatre, the surgical waste is destroyed.
  Instead of being destroyed, the leg will be used for research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: artericitc surgery — biological sample (leg) from leg amputation surgery used for research

SUMMARY:
PRIMARY OBJECTIVE Qualitatively describe the distribution of cutaneous arteries in patients with long-term occlusive arterial disease.

SECONDARY OBJECTIVE To compare the distribution of cutaneous arteries observed on the legs of arteritic patients with that observed on non-arteritic legs (from bodies given to science).

DETAILED DESCRIPTION:
Arterial patient coming to CHRU Nancy, in the Vascular and Endoluminal Surgery Department, to undergo leg amputation.

Usually, after the amputation of the leg in the operating theatre, the surgical waste is destroyed.

Instead of being destroyed, the leg will be used for research.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Patient with late stage occlusive arteriopathy with lower limb amputation
* Patient who did not oppose the search
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients with infectious diseases not accessible in the anatomy laboratory
* Woman of childbearing age without effective contraception
* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code :
* Pregnant woman, parturient or nursing mother
* Person deprived of liberty by a judicial or administrative decision,
* Person under psychiatric care pursuant to Articles L.3212-1 and L.3213-1 of the Public Health Code
* Person admitted to a health or social institution for purposes other than research
* Minor person (not emancipated)
* Adult subject to a legal protection measure (guardianship, trusteeship, protection of justice)
* Major person who is not in a position to express consent and who is not subject to a legal protection measure

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: arteritic patient coming to CHRUN as part of the care
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative mapping of the skin's arteries. | 72 hours after the dissection of the leg.
  The leg will be transported in a container to the Anatomy Laboratory (Faculty of Medicine - University of Lorraine).
  Within 72 hours of its arrival, the operating room will be dissected to qualitatively describe the distribution of cutaneous arteries in patients with long-term occlusive arterial disease.